CLINICAL TRIAL: NCT03408587
Title: An Open-Label Phase 1b Clinical Study of Intravenous CAVATAK® (Coxsackievirus A21, CVA21), in Combination With Ipilimumab in Subjects With Uveal Melanoma Metastatic to Liver (VLA-024 CLEVER)
Brief Title: CAVATAK® and Ipilimumab in Uveal Melanoma Metastatic to the Liver (VLA-024 CLEVER)
Acronym: CLEVER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viralytics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V937-010; VLA-024 (Other: Viralytics Study ID)
Record Dates: First submitted 2018-01-10; First posted 2018-01-24 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Uveal Melanoma; Liver Metastases
Keywords: CVA21; CAVATAK; Coxsackievirus; ocular; eye; ipilimumab; yervoy; oncolytic; virus; checkpoint; CTLA-4
MeSH Terms: conditions — Uveal Melanoma; Coxsackievirus Infections; Virus Diseases; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Ipilimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CVA21 / Ipilimumab (Experimental): Subjects will receive up to 8 cycles (Day 155) of intravenous CVA21 and 4 doses of ipilimumab (Days 8, 29, 50 and 71).
  Interventions: Biological: CVA21; Biological: Ipilimumab

INTERVENTIONS:
Biological: CVA21 — Oncolytic virus
  Other Names: CAVATAK, Coxsackievirus A21
Biological: Ipilimumab — Fully human IgG1 monoclonal antibody that binds to the CTLA-4 receptor expressed on activated T cells.
  Other Names: Yervoy

SUMMARY:
This is an open-label Phase 1b clinical study of ipilimumab in combination with intravenous CVA21 in subjects who have uveal melanoma metastatic to liver.

DETAILED DESCRIPTION:
This is an open-label Phase 1b clinical study of ipilimumab in combination with intravenous CVA21 in subjects who have uveal melanoma metastatic to liver. Subjects will receive up to 8 cycles of CVA21 at a planned dose of 1 x 10e9 TCID50 per infusion, with the first cycle being a 28-day cycle consisting of an intravenous infusion on Days 1, 3, 5 and 8 and subsequent cycles every 21 days from Day 8.

Ipilimumab will be given by intravenous administration at a dose of 3mg/kg, for a maximum of 4 doses, given on Days 8, 29, 50 and 71. On days when both CVA21 and ipilimumab are given, CVA21 will be given first.

Subjects will be monitored for treatment toxicity using the current version of CTCAE.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologically confirmed diagnosis of uveal melanoma with measurable disease (based on RECIST 1.1 criteria) in the liver (by CT, PET/CT or MRI) at the time of screening.
2. Patients that have had prior treatment must show disease progression during or following the last treatment according to RECIST 1.1 criteria.
3. Men and women ≥ 18 years of age.
4. The subject has a life expectancy of greater than 12 weeks.
5. The subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Adequate organ function as defined by and obtained within 28 days of starting treatment:

   * Absolute neutrophil count ≥ 1,500 /mcl
   * WBC ≥ 3.0 x 10e9/L
   * Platelets ≥ 100,000 /mcl
   * Hemoglobin ≥ 9 g/dL
   * Creatinine ≤ 1.5 x ULN
   * Albumin > 3 g/dL
   * Total bilirubin ≤ 1.5 x ULN or direct bilirubin ≤ ULN for subjects with total bilirubin > 1.5 x ULN
   * AST and ALT ≤ 5 x ULN
   * INR or PT ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT and PTT are within therapeutic range of intended use of anticoagulants.
   * aPTT ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT and PTT are within therapeutic range of intended use of anticoagulants.
7. Prior therapy with an immune checkpoint inhibitor therapy is allowable. A 6-week washout period will be required for those with prior PD-1 or PD-L1 treatment.
8. Female subjects of child-bearing potential must have a negative urine pregnancy test within 72 hours prior to receiving the first dose of study medication. If a urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female and Male subjects of childbearing potential must be willing to use an adequate method of contraception, starting with the first dose of study drug through 4 weeks after the last dose of study drug. Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
10. The subject is capable of understanding and complying with protocol requirements.
11. The subject or the subject's legally acceptable representative provides written, informed consent prior to the initiation of any study procedures.

Exclusion Criteria:

1. The subject is a candidate for surgery or loco-regional treatment with curative intent.
2. Subjects with active (i.e. symptomatic or growing) central nervous system (CNS) metastases. Subjects with CNS metastases are eligible if the metastases have been treated with surgery and/or radiotherapy, the subject is off corticosteroids for at least 2 weeks and the subject is neurologically stable.
3. Known additional malignancy that is progressing or requires active treatment. Exceptions include cutaneous squamous cell or basal cell carcinoma that has undergone potentially curative therapy or in-situ cervical cancer.
4. Known history of Human Immunodeficiency Virus (HIV, HIV 1/2 antibodies), known active Hepatitis B (e.g. HBsAg reactive) or Hepatitis C (e.g. HCV RNA [qualitative] is detected).
5. Current systemic steroid therapy other than physiologic replacement (i.e. prednisone ≤ 10 mg or equivalent). Inhaled or topical steroid use is allowed.
6. Active auto-immune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.
7. Active colitis or previous immune-mediated colitis that has not resolved to grade 1 or less.
8. Chemotherapy, targeted small molecule therapy, radiation therapy, hormonal treatment or immunotherapy within 21 days prior to initiation of treatment. A 6-week washout period will be required for those with prior PD-1 or PD-L1 treatment. Subjects must have resolution of toxic effect(s) of the most recent therapy to Grade 1 or less. Exceptions are subjects with ≤ Grade 2 alopecia or ≤ Grade 2 neuropathy who are permitted in the study. If the subject received major surgery or radiation therapy of >30 Gy, they must have recovered from the toxicity and/or any complications from the intervention.
9. Pregnancy, breastfeeding, or expectation to conceive or father children within the projected duration of the trial, starting with the screening visit through 4 weeks after the last dose of study treatment.
10. Known sensitivity to any of the products or components to be administered during dosing.
11. Participation in a study of an investigational agent or device within 4 weeks of Day 1.
12. Subjects with any other concurrent, uncontrolled illness, including known psychiatric or substance abuse disorders which may interfere with the ability of the subject to cooperate and participate in the trial. Other examples of such conditions would include unstable angina, myocardial infarction (MI) or cerebrovascular accident (CVA) within 6 months of study entry.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Patients with tumors lying close to an airway, major blood vessel or spinal cord that, in the opinion of the investigator, could cause occlusion or compression in the case of swelling, or erosion into a major vessel in the case of necrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events as assessed using the current NCI-CTCAE. | 30 days from the last administration of study treatment
  Treatment-emergent adverse events (TEAEs) are defined as AEs that start on or after the first day of study treatment and within 30 days of the last administration of study treatment. The incidence of TEAEs will be summarized based on the number and percentage of subjects who experience events classified by MedDRA system organ class and preferred term.

SECONDARY OUTCOMES:
Overall Response Rate | 2 years
  Objective responses will be assessed according to immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jose Lutzky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Lutzky J, Sullivan RJ, Cohen JV, Ren Y, Li A, Haq R. Phase 1b study of intravenous coxsackievirus A21 (V937) and ipilimumab for patients with metastatic uveal melanoma. J Cancer Res Clin Oncol. 2023 Aug;149(9):6059-6066. doi: 10.1007/s00432-022-04510-3. Epub 2023 Jan 18. PMID 36651961